CLINICAL TRIAL: NCT01743001
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Phase 3 Study to Evaluate the Effects of Macitentan on Exercise Capacity in Subjects With Eisenmenger Syndrome
Brief Title: Clinical Study to Evaluate the Effects of Macitentan on Exercise Capacity in Subjects With Eisenmenger Syndrome
Acronym: MAESTRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055-305
Record Dates: First submitted 2012-11-29; First posted 2012-12-06 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: exercise capacity; Eisenmenger Syndrome
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Eisenmenger Complex | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Macitentan (Experimental): Subjects receive macitentan 10 mg oral tablet once daily
  Interventions: Drug: Macitentan 10 mg
- Placebo (Placebo Comparator): Subjects receive macitentan-matching placebo oral tablet once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macitentan 10 mg — Macitentan 10 mg oral tablet once daily
  Other Names: ACT-064992
  Arms: Macitentan
Drug: Placebo — Macitentan-matching placebo oral tablet once daily
  Arms: Placebo

SUMMARY:
Clinical study to assess the efficacy, safety, and tolerability of macitentan in subjects with Eisenmenger Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects:

  * not participating in the hemodynamic sub-study: males or females ≥ 12 years of age.
  * participating in the hemodynamic sub-study: males or females ≥ 18 years of age.
* Subjects (including those with Down Syndrome [DS]) with confirmed Eisenmenger Syndrome [ES] (European Society of Cardiology [ESC] and the European Respiratory Society [ERS] guidelines):

  1. Established by echocardiography as:

     * Large congenital shunting defect at atrial, ventricular or arterial level*
     * and right to left shunt or bi-directional shunt with prevalent right to left direction.
  2. Resting peripheral oxygen saturation (SpO2) ≤ 90% and > 70% (pulse oximetry, room air).

The lower limit is 65% if a subject is living at an altitude greater than 2500 m above sea level.

*Subjects with any of the following open defects are eligible for the study either as an isolated defect or in combination:

* atrial septal defect (ASD)
* ventricular septal defect (VSD)
* partial or complete atrioventricular septal defect (AVSD)
* patent ductus arteriosus (PDA)
* aortopulmonary window (AP window)
* total or partial anomalous pulmonary venous return (TAPVR, PAPVR) The defects may be either unoperated or previously palliated surgically (provided significant residual defect remains).

The Steering Committee will review the echocardiography data of all subjects (main study and sub study) to confirm eligibility prior to Randomization.

* Subjects with the following findings at cardiac catheterization:

  * Mean resting pulmonary arterial pressure (mPAP) > 25 mmHg
  * Pulmonary capillary wedge pressure (PCWP) or mean left atrial pressure (LAP) or left ventricular end diastolic pressure (LVED) ≤ 15 mmHg
  * Pulmonary vascular resistance (PVR) ≥ 800 dyn∙s/cm5 or ≥ 10 Wood units
* Subjects with WHO functional class ≥ II.
* Subjects able to reliably perform the the 6-minute walk test (6MWT) with a minimum distance of 50 m and a maximum distance of 450 m.

Exclusion Criteria:

- Main study and hemodynamic sub-study: Any of the following conditions previously known or identified via cardiac catheterization or echocardiography:

* Pulmonary arterial or venous stenosis > 25% size of native pulmonary artery (PA) or pulmonary vein
* Severe tricuspid regurgitation in the setting of left to right shunt at the ventricular or atrial level
* Greater than mild tricuspid stenosis
* Intracavitary RV outflow obstruction
* Greater than mild mitral stenosis
* Intracavitary LV outflow obstruction
* Subvalvular or supravalvular aortic stenosis
* Aortic coarctation
* Greater than moderate mitral regurgitation
* Recognized extracardiac systemic venous collaterals to the pulmonary venous circulation
* Recognized hepatic wedge pressure-inferior vena cava pressure gradient >12 mm Hg
* PCWP "v" waves >20 mmHg
* Tetralogy of Fallot
* Truncus arteriosus
* Interrupted aortic arch
* Transposition of great arteries
* Single ventricle defects: absent AV connection (mitral or tricuspid atresia), double inlet AV connections left or right ventricle, functional univentricular heart (unbalanced AVSD, hypoplastic RV, double outlet RV), hypoplastic left heart syndrome
* Ebstein's anomaly
* Severe aortic regurgitation
* Pulmonary atresia
* PAPVR or TAPVR, ONLY if there is lung hypoplasia or if documentation confirming the absence of lung hypoplasia does not exist.

For subjects participating in the hemodynamic sub-study the following will also be considered exclusion criteria:

* SVC stenosis >25% size of native vessel
* PDA, AP window, TAPVR, PAPVR, or ASD sinus venosus with anomalous pulmonary veins
* Down Syndrome

  * Subjects with deterioration of their clinical status within 3 months prior to Screening or during the Screening period.
  * Known moderate-to-severe restrictive (i.e., total lung capacity [TLC] < 60% of predicted value) or obstructive lung disease (i.e., forced expiratory volume in one second [FEV1] < 80 % of predicted value, and with FEV1 / forced vital capacity [FVC] < 70%)
  * Treatment with prostanoids within 1 month prior to Randomization
  * Subjects who initiated a PDE-5 inhibitor within 1 month prior to Randomization or those on a PDE-5 inhibitor for whom the dose has not been stable within 1 month prior to Randomization
  * Treatment with endothelin receptor antagonists (ERAs) within 1 month prior to Randomization
  * Subjects who initiated diuretics within 1 week prior to Randomization or subjects whose diuretic treatment has not been stable for at least 1 week prior to Randomization
  * Subjects being considered for an organ transplant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (7):
  - Ahmanson/UCLA Heart Disease Center, Los Angeles, California
  - Stanford Hospital and Clinic, Palo Alto, California
  - Emory University Hospital/the Emory Clinic, Atlanta, Georgia
  - Barnes-Jewish Hosp/Wash Univ School of Med, St Louis, Missouri
  - Children'S Heart Center Nevada, Las Vegas, Nevada
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Children'S Hosp - Dept of Cardiology, Houston, Texas
- Gen Hosp Univ Vienna Dept Cardiology, Vienna, Austria
- Bulgaria (3):
  - Mhat Nat Card Hosp - Cardiology Clinic, Sofia
  - Mhat Nat Card Hosp - Pediatric Clin / Ped Card Dept, Sofia
  - Mhat Sveta Anna Clin Card, Sofia
- Chile (2):
  - Inst Nat Torax, Unidad Cardiopatia Congenitas Del Adulto, Providencia
  - Clinica Tabancura - Cardio Unit, Santiago
- China (6):
  - Guangdong General Hospital, Cardiology Dpt, Guangzhou, Guangdong
  - Wu Han Asia Heart Hosp, Wuhan, Hubei
  - The General Hosp of Shenyang Military Region, Shenyang, Liaoning
  - Beijing Anzhen Hospital, Cardiology Dpt, Beijing
  - Cardiovascular Institute&Fuwai Hospital, Beijing
  - Shanghai Pulmonary Hospital, Dept of Pulmonary Circulation, Shanghai
- France (4):
  - Hosp La Timone - Dept Pediatric Cardiology, Marseille
  - Hosp Laennec - Dept Cardiology, Nantes
  - Hosp Pompidou - Dept Congenital Cardiac Diseases, Paris
  - Hosp Cardiology Haut Leveque - Dept Congenital Diseases, Pessac
- Germany (3):
  - Herzzentrum Berlin, Ped Cardiology, Berlin
  - Universitätsklinikum Giessen - Pediatric Heart Center, Giessen
  - Uni Heidelberg - Kinderkardiologie, Heidelberg
- Ahepa University General Hospital, Thessaloniki, Greece
- Rabin Medical Centre - Pulmonology, Petach Tikvah, Israel
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Mexico (3):
  - Unidad de Investigacion Clin En Med, Sc (Udicem), Monterrey, Nuevo León
  - Instituto Nacional de Cardiologia (Inc) Ignacio Chavez, Mexico City
  - Instituto de Corazon de Querètaro, Querétaro
- PHC, MAB, Manila, Philippines
- Poland (3):
  - Cardiology Gdańsk Univ, Gdansk
  - Cardiology Kraków Univ, Krakow
  - Cardiology Wrocław, Wroclaw
- Portugal (2):
  - Hosp Univ Coimbra - Dpt Cardiology, Coimbra
  - Hosp Sta Marta - Dept Cardiology, Lisbon
- Romania (3):
  - Er Inst For Cardvasc Dis "Prof Dr Cc Iliescu" - Card Ii, Bucharest
  - Cardio Med Srl, Târgu Mureş
  - Clin Hosp For Inf and Pulm Dis Victor Babes - Ii Pulm, Timișoara
- Russia (3):
  - Sci Institute Systemic Problems Cardio Diseases Kemerovo, Kemerovo
  - Russian Cardiology Scientific and Production Complex, Moscow
  - V. A. Almazov Institute of Cardiology, Saint Petersburg
- Serbia (3):
  - Dedinje Cardiovasc Inst - Cardiovasc Research Ctr, Belgrade
  - Mother and Child Health Care Inst "Dr Vukan Cupic", Belgrade
  - Clin Hosp Ctr Zemun - Cardiology Dept, Belgrade
- Spain (3):
  - Hosp Univ Vall D'Hebron - Dpt Congenital Heart Disease Adult, Barcelona
  - Hosp Univ Virgen Macarena - Dpt Cardiology, Seville
  - Hosp Universitario La Fe Dpt Cardiology, Valencia
- Omu Pediatry, Samsun, Turkey (Türkiye)
- Bristol Univ Hosp Congenital Heart Centre, Bristol, United Kingdom
- Vietnam (3):
  - Hanoi Medical University Hospital, Hanoi
  - Children's Hospital, Ho Chi Minh, Ho Chi Minh City
  - Tam Duc Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Gatzoulis MA, Landzberg M, Beghetti M, Berger RM, Efficace M, Gesang S, He J, Papadakis K, Pulido T, Galie N; MAESTRO Study Investigators. Evaluation of Macitentan in Patients With Eisenmenger Syndrome. Circulation. 2019 Jan 2;139(1):51-63. doi: 10.1161/CIRCULATIONAHA.118.033575. PMID 30586694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 71 sites in 26 countries (geographical regions: Asia-Pacific, Eastern Europe, Latin America, North America, Western Europe including Israel and Turkey, and South Africa), of which 55 sites in 21 countries randomized subjects.
Pre-assignment Details: The screening period lasted a maximum of 30 days from Visit 1 up to Randomization (Visit 2). A total of 319 subjects were screened and 226 subjects were randomized to macitentan 10 mg and placebo.
Groups:
- Macitentan: Subjects receive macitentan 10 mg, oral tablet, to be taken once daily
- Placebo: Subjects receive macitentan-matching placebo, oral tablet, to be taken once daily
Period: Overall Study
Arm/Group | Macitentan | Placebo
Started | 114 | 112
Completed | 111 | 112
Not Completed | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan | Placebo | Total
Number analyzed (Participants) | 114 | 112 | 226
Age, Continuous [Median (Full Range); unit: Years] | 33.0 [12 to 82] | 31.0 [13 to 62] | 32.0 [12 to 82]
Age, Customized [Count of Participants; unit: Participants]
  12 - 17 years | 13 | 2 | 15
  18 - 55 years | 90 | 105 | 195
  ≥ 56 years | 11 | 5 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 68 | 150
  Male | 32 | 44 | 76
Region of Enrollment [Count of Participants; unit: Participants] — Asia-Pacific includes: China, Malaysia, Philippines, Vietnam; Eastern Europe: Bulgaria, Poland, Romania, Russian Federation, Serbia; Latin America: Chile, Mexico; North America: United States; Western Europe - Israel: Austria, France, Germany, Greece, Israel, Portugal, Spain, Turkey, United Kingdom
  Participants
    Asia-Pacific | 47 | 44 | 91
    Eastern Europe | 25 | 27 | 52
    Latin America | 19 | 18 | 37
    North America | 2 | 5 | 7
    Western Europe - Israel | 21 | 18 | 39
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 21.15 [11.9 to 38.9] | 21.55 [14.5 to 42.2] | 21.35 [11.9 to 42.2]
WHO functional class [Count of Participants; unit: Participants] — Class I: no symptoms with exercise or at rest. No limitation of activity. Class II: No symptoms at rest but slight limitation with ordinary activities causing symptoms (e.g. short of breath with climbing a flight of stairs, grocery shopping, or making the bed). Class III: may not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. Class IV: symptoms at rest (e.g. dyspnea and/or fatigue) and inability to carry out any physical activity without symptoms. Patients in class IV manifest signs of right heart failure. Population: Per protocol patients in WHO functional class I were excluded.
  Participants
    class I | 0 | 0 | 0
    class II | 69 | 66 | 135
    class III | 45 | 46 | 91
    class IV | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in Exercise Capacity, as Measured by 6-minute Walk Distance (6MWD)
Description: The purpose of the six minute walk is to test exercise tolerance and capacity. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Frame: From baseline to Week 16
Population: Full analysis set: The analysis was performed on the full analysis set (FAS), i.e., all randomized subjects in the treatment group to which they were randomized and by imputing missing values at Week 16 according to pre-defined rules.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 114 | 112
meter
  6MWD at baseline | 368.7 (74.5) | 380.3 (76.3)
  6MWD at Week 16 | 387.1 (101.8) | 399.9 (79.5)
  Change in 6MWD from baseline to Week 16 | 18.3 (84.4) | 19.7 (53.0)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The null hypothesis was that there was no difference between macitentan and placebo for the mean change from baseline to Week 16 in 6MWD. Null hypothesis was tested by an analysis of covariance (ANCOVA); Test type: Superiority; p = 0.6120, ANCOVA — To control for multiplicity across the primary and secondary endpoints, all secondary endpoints were analyzed hierarchically according to order and significance as pre-specified in the protocol eliminating further adjustment for multiple comparisons; ANCOVA model included treatment group, presence of DS (yes/no), and WHO FC (II vs III/IV) as categorical factors, and baseline 6MWD value as covariate; least-square (LS) mean difference = -4.7, 95% CI 2-sided [-22.8 to 13.5]

2. Secondary Outcome: Change From Baseline to Week 16 in WHO Functional Class
Description: A shift in WHO functional classes is considered an 'improvement' when shifting to a lower class (e.g. from class III to class II) or a 'worsening' when shifting to a higher class (e.g. from class III to class IV). Definition of functional classes as follows - Class I: no symptoms with exercise or at rest. Class II: No symptoms at rest but uncomfortable and short of breath with normal activity such as climbing a flight of stairs, grocery shopping, or making the bed. Class III: May not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting (e.g. doing normal chores around the house, have to take breaks while doing activities of daily living). Class IV: Symptoms at rest and severe symptoms with any activity. Most patients also have edema in the feet and ankles as result of right heart failure.
Time Frame: From baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 114 | 112
Participants
  WHO functional class 1 at Week 16 | 3 | 1
  WHO functional class 2 at Week 16 | 72 | 79
  WHO functional class 3 at Week 16 | 38 | 32
  WHO functional class 4 at Week 16 | 1 | 0
  Unchanged from baseline to Week 16 | 103 | 95
  Improvement from baseline to Week 16 | 10 | 16
  Worsening from baseline to Week 16 | 1 | 1
Statistical Analysis 1: Comparison: Macitentan vs Placebo; For this secondary endpoint of WHO functional class, the improvement from baseline to Week 16 in WHO functional class was evaluated. The null hypothesis is the odds of improvement are the same in the placebo and the macitentan group; Test type: Superiority; p = 0.1450, Regression, Logistic — The secondary efficacy endpoints were analyzed hierarchically as this approach eliminated the requirement for further adjustment for multiple comparisons; Logistic regression model adjusted for randomized treatment group and location of cardiac defect (pre-tricupsid / post-tricupsid ) as factors; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.23 to 1.24]

3. Secondary Outcome: Change From Baseline to Week 16 in Dyspnea, Assessed by the Borg Dyspnea Index
Description: This outcome measures the difference in the Borg dyspnea index collected at the end of the 6-minute walk test (6MWT) at Week 16 compared to baseline. The Borg dyspnea index rates the severity of dyspnea (difficult or labored breathing) on a scale from 0 ('Nothing at all') to 10 ('Very, very severe - maximal'). A decrease in the Borg dyspnea index indicates an improvement.
Time Frame: From baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 114 | 112
Score on a scale
  Borg dyspnea index score at baseline | 3.00 (1.95) | 2.94 (1.88)
  Borg dyspnea index score at Week 16 | 2.78 (2.10) | 2.66 (1.64)
  Change from baseline to Week 16 | -0.22 (1.56) | -0.29 (1.50)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The null hypothesis was that the mean change from baseline to Week 16 in the Borg dyspnea index is the same in the macitentan and in the placebo group; Test type: Superiority; p = 0.6818, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted for randomized treatment group, location of cardiac defect(pre-tricupsid/post-tricupsid) as factors, baseline Borg dyspnea index as covariate; least-square (LS) mean difference = 0.08, 95% CI [-0.29 to 0.44]

4. Secondary Outcome: Change From Baseline to Week 16 in Quality of Life (QoL), Assessed by the Short Form-36 (SF-36) Questionnaire
Description: The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of the functional health and well-being scores (i.e., physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health), as well as psychometrically based physical and mental health summary measures and a preference-based health utility (health rated as much better now than one year ago to much worse now than one year ago). It is a generic measure, as opposed to one that targets a specific age, disease, or treatment group.
  For each of the domains and scores that the SF36 measures an aggregate percentage score is produced. The percentage scores range from 0% (lowest or worst possible level of functioning) to 100% (highest or best possible level of functioning). A higher score for the individual domains and summary component scores indicates a better condition of the subject.
Time Frame: From baseline to Week 16
Population: Full analysis set (excluding children <14 years of age and Down Syndrome subjects)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 101 | 99
Score on a scale
  Domain score: physical functioning at baseline | 51.9 (21.8) | 52.7 (22.4)
  Domain score: physical functioning at Week 16 | 56.4 (21.9) | 58.0 (19.7)
  Change in physical functioning (domain score) | 4.6 (16.5) | 5.3 (15.4)
  Domain score: role-physical at baseline | 46.2 (25.5) | 48.4 (27.9)
  Domain score: role-physical at Week 16 | 52.8 (25.5) | 55.9 (25.3)
  Change in role-physical (domain score) | 6.6 (20.1) | 7.4 (22.1)
  Domain score: pain index at baseline | 61.7 (23.0) | 64.6 (24.6)
  Domain score: pain index at Week 16 | 65.2 (23.6) | 66.2 (24.7)
  Change in pain index (domain score) | 3.5 (22.1) | 1.6 (27.1)
  Domain score:general health perceptions baseline | 36.1 (21.0) | 37.2 (19.8)
  Domain score:general health perceptions at Week 16 | 40.3 (22.7) | 37.6 (20.3)
  Change in general health perceptions(domain score) | 4.2 (16.4) | 0.5 (15.5)
  Domain score: vitality at baseline | 49.0 (22.1) | 51.9 (21.5)
  Domain score: vitality at Week 16 | 56.1 (19.8) | 56.3 (17.5)
  Change in vitality (domain score) | 7.1 (18.3) | 4.4 (18.2)
  Domain score: social functioning at baseline | 64.7 (26.8) | 66.9 (25.0)
  Domain score: social functioning at Week 16 | 66.6 (25.8) | 69.2 (23.5)
  Change in social functioning (domain score) | 1.9 (23.0) | 2.3 (24.5)
  Domain score: role-emotional at baseline | 61.6 (27.4) | 61.3 (28.8)
  Domain score: role-emotional at Week 16 | 63.3 (26.8) | 66.0 (25.6)
  Change in role-emotional (domain score) | 1.7 (22.8) | 4.7 (25.0)
  Domain score: mental health index at baseline | 63.8 (21.1) | 64.0 (20.5)
  Domain score: mental health index at Week 16 | 65.7 (18.9) | 67.7 (20.6)
  Change in mental health index (domain score) | 1.9 (16.1) | 3.7 (16.6)
  Norm-based: physical functioning at baseline | 36.8 (9.2) | 37.1 (9.4)
  Norm-based: physical functioning at Week 16 | 38.7 (9.2) | 39.3 (8.3)
  Change in physical functioning (norm-based) | 1.9 (6.9) | 2.2 (6.5)
  Norm-based: role-physical at baseline | 35.8 (10.0) | 36.6 (10.9)
  Norm-based: role-physical at Week 16 | 38.4 (10.0) | 39.6 (9.9)
  Change in role-physical (norm-based) | 2.6 (7.9) | 2.9 (8.7)
  Norm-based: pain index at baseline | 45.9 (9.7) | 47.2 (10.4)
  Norm-based: pain index at Week 16 | 47.4 (10.0) | 47.8 (10.4)
  Change in pain index (norm-based) | 1.5 (9.3) | 0.7 (11.5)
  Norm-based: general health perceptions at baseline | 33.4 (10.0) | 33.9 (9.4)
  Norm-based: general health perceptions at Week 16 | 35.4 (10.8) | 34.2 (9.7)
  Change in general health perceptions (norm-based) | 2.0 (7.8) | 0.2 (7.4)
  Norm-based: vitality at baseline | 45.4 (11.1) | 46.8 (10.7)
  Norm-based: vitality at Week 16 | 48.9 (9.9) | 49.0 (8.7)
  Change in vitality (norm-based) | 3.6 (9.1) | 2.2 (9.1)
  Norm-based: social functioning at baseline | 41.5 (11.7) | 42.4 (10.9)
  Norm-based: social functioning at Week 16 | 42.3 (11.3) | 43.4 (10.3)
  Change in social functioning (norm-based) | 0.8 (10.0) | 1.0 (10.7)
  Norm-based: role-emotional at baseline | 37.9 (12.8) | 37.8 (13.4)
  Norm-based: role-emotional at Week 16 | 38.8 (12.5) | 40.0 (11.9)
  Change in role-emotional (norm-based) | 0.8 (10.6) | 2.2 (11.7)
  Norm-based: mental health index at baseline | 43.7 (11.9) | 43.8 (11.6)
  Norm-based: mental health index at Week 16 | 44.8 (10.6) | 45.9 (11.6)
  Change in mental health index (norm-based) | 1.1 (9.1) | 2.1 (9.3)
  Physical component summary score at baseline | 37.6 (7.5) | 38.6 (8.7)
  Physical component summary score at Week 16 | 40.0 (8.4) | 40.0 (7.7)
  Change in physical component summary score | 2.4 (6.4) | 1.4 (6.5)
  Mental component summary score at baseline | 43.8 (12.4) | 44.1 (12.1)
  Mental component summary score at Week 16 | 44.7 (11.7) | 45.9 (10.9)
  Change in mental component summary score | 1.0 (9.3) | 1.8 (9.3)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Physical Functioning; Test type: Superiority; p = 0.6431, ANCOVA; Adjusted for randomized treatment group, location of cardiac defect (pre-tricupsid/post-tricupsid) as factors and baseline scores as covariates; least-square (LS) mean difference = -1.0, 95% CI 2-sided [-5.0 to 3.1]
Statistical Analysis 2: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Role-Physical; Test type: Superiority; p = 0.5988, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -1.4, 95% CI 2-sided [-6.7 to 3.9]
Statistical Analysis 3: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Pain Index; Test type: Superiority; p = 0.9642, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = 0.1, 95% CI 2-sided [-5.9 to 6.2]
Statistical Analysis 4: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of General Health Perceptions; Test type: Superiority; p = 0.1542, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = 3.1, 95% CI 2-sided [-1.2 to 7.3]
Statistical Analysis 5: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Vitality; Test type: Superiority; p = 0.6020, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = 1.1, 95% CI 2-sided [-3.1 to 5.3]
Statistical Analysis 6: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Social Functioning; Test type: Superiority; p = 0.6340, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -1.4, 95% CI 2-sided [-7.2 to 4.4]
Statistical Analysis 7: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Role-Emotional; Test type: Superiority; p = 0.3384, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -2.8, 95% CI 2-sided [-8.7 to 3.0]
Statistical Analysis 8: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Mental Health Index; Test type: Superiority; p = 0.2704, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -2.3, 95% CI 2-sided [-6.4 to 1.8]
Statistical Analysis 9: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Physical Functioning (norm-based); Test type: Superiority; p = 0.6431, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -0.4, 95% CI 2-sided [-2.1 to 1.3]
Statistical Analysis 10: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Role-Physical (norm-based); Test type: Superiority; p = 0.5988, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -0.6, 95% CI 2-sided [-2.6 to 1.5]
Statistical Analysis 11: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Pain Index (norm-based); Test type: Superiority; p = 0.9642, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = 0.1, 95% CI 2-sided [-2.5 to 2.6]
Statistical Analysis 12: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of General Health Perceptions (norm-based); Test type: Superiority; p = 0.1542, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = 1.5, 95% CI 2-sided [-0.6 to 3.5]
Statistical Analysis 13: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Vitality (norm-based); Test type: Superiority; p = 0.6020, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = 0.6, 95% CI 2-sided [-1.5 to 2.6]
Statistical Analysis 14: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Social Functioning (norm-based); Test type: Superiority; p = 0.6340, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -0.6, 95% CI 2-sided [-3.1 to 1.9]
Statistical Analysis 15: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the SF-36 domain score of Role-Emotional (norm-based); Test type: Superiority; p = 0.3384, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -1.3, 95% CI 2-sided [-4.1 to 1.4]
Statistical Analysis 16: Comparison: Macitentan vs Placebo; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.2704, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -1.3, 95% CI 2-sided [-3.6 to 1.0]
Statistical Analysis 17: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the Physical Component Summary Score; Test type: Superiority; p = 0.4332, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = 0.7, 95% CI 2-sided [-1.0 to 2.3]
Statistical Analysis 18: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline to Week 16 is the same in the macitentan and the placebo group for the Mental Component Summary Score; Test type: Superiority; p = 0.3416, ANCOVA; [statistical method as in outcome 4, analysis 1]; least-square (LS) mean difference = -1.1, 95% CI 2-sided [-3.4 to 1.2]

ADVERSE EVENTS:
Time Frame: A safety follow-up visit was required 30 days after end of treatment period at Week 16. Subjects who prematurely discontinued treatment prior to Week 16 were required to perform a premature end-of-treatment visit no later than 7 days after last dose of study treatment and then followed by the 30 day safety follow-up visit.
Groups:
- Macitentan: Subjects receive macitentan 10 mg orally to be taken once daily. 114 subjects were exposed to Macitentan 10 mg for 15.93 weeks on average.
- Placebo: Subjects receive macitentan-matching placebo orally to be taken once daily. 112 subjects were exposed to placebo for 15.96 weeks on average.
Arm/Group | Macitentan | Placebo
All-Cause Mortality (participants affected / at risk) | 1/114 | 0/112
Serious Adverse Events (participants affected / at risk) | 7/114 | 2/112
Other Adverse Events (participants affected / at risk) | 31/114 | 30/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=114) | Placebo (N=112)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 3 (4) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=114) | Placebo (N=112)
Bronchitis (Infections and infestations) | 6 (6) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (8)
Headache (Nervous system disorders) | 13 (15) | 5 (5)
Nasopharyngitis (Infections and infestations) | 3 (4) | 14 (16)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 60 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.